CLINICAL TRIAL: NCT03979924
Title: Trismus Prevalence and Preventive Rehabilitation Associated With Therapeutic Education for Patients With Head and Neck Cancer Treated With Concomitant Radiochemotherapy
Brief Title: Mouth Opening, Prevention, Education, Nutrition (OPEN)
Acronym: OPEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICM-URC 2016-08
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Trismus; Head and Neck Cancer
Keywords: Trismus; prevention; education; nutrition; preventive rehabilitation; mouth
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Step (Other): The interventional step will comprise the same follow-up as the observational step, except for the addition of an early and preventive care, conducted by a specialized physiotherapist using an active exercise handbook elaborated with the patient's therapeutic education transversal Unit (Utep). This aims at increasing the patient's adhesion to the program and to limit the reduction of mouth opening and its consequences ( Trismus rehabilitation)
  Interventions: Behavioral: Trismus rehabilitation

INTERVENTIONS:
Behavioral: Trismus rehabilitation — The patient will be followed-up by a physiotherapist during all the whole radiotherapy treatment, with short 15-min sessions, twice a week. He/she will be trained to perform regularly and by him/herself the preventive/rehabilitation exercises than the patient will do twice a day until the end of the radiotherapy treatment. The patient will then continue, in an autonomous manner, with his/her rehabilitation.
  In case of trismus occurrence, the physiotherapist will advise the patient to add a passive tool to the active exercises (Jaw Trainer, Therabite, tongue depressors,…) in order to strengthen the stretching.

SUMMARY:
In France, 11 316 new cases of upper aero-digestive tract cancer were estimated in 2012. These cancers are treated with a triple-therapy combining surgery, radiotherapy and chemotherapy/targeted therapies. Treatment-induced sequelae are often burdensome: reduction in mouth opening, eventually on to trismus, limitation of lips and tongue mobility, deterioration in oral hygiene, pain due to inflammation and muscle fibrosis. Trismus is defined as a mouth opening of less than 35mm in patients with head and neck cancers. It can be induced by treatments (surgery or radiotherapy) but is also reported at the time of diagnosis, due to the local evolution of the tumour.

Management of trismus and its consequences is currently mostly based on physiotherapy of maxillary constrictions in order to limit or decrease the reduction of mouth opening in these patients. Exercise protocols have been set up and evaluated in the literature, but with various results. The benefit of a physiotherapy intervention on trismus prevalence, mouth opening, and patients' quality of life has not yet been shown.

Our hypothesis is that at least 30% of patients treated with radiochemotherapy are affected by trismus. According to the nutrition national recommendations in oncology, patients the most at-risk of loco-regional complications are those who receive radiotherapy doses of 54Gy or more in the oropharynx and concomitant chemotherapy.

It is thus essential to provide these patients with an early and preventive management of trismus and its consequences, during the whole duration of the treatment.

DETAILED DESCRIPTION:
The management of trismus and its side effects is essentially based on a re-education of maxillary constrictions to limit or reduce the loss of mouth opening in patients. Exercise protocols are in place and have been evaluated in the literature with discordant results. The beneficial effect of a rehabilitation program on the prevalence of trismus, oral opening and quality of life of patients is not yet clearly demonstrated.

Three studies did not show any significant beneficial effect of rehabilitation programs nor on the prevalence of trismus or the quality of life of patients. A 2014 randomized trial showed no benefit from a passive exercise program on trismus prevention and oral opening. Another 2011 study compared 374 patients, a control group and an intervention group following language mobility exercises, rehabilitation supervised by a physiotherapist and specific trismus prevention exercises with the help of a doctor. specific tool (Jaw Trainer) during and after radiotherapy. A third, more recent, randomized study evaluated the effect of a very comprehensive rehabilitation program consisting of a 45-minute session per week of rehabilitation with a physiotherapist, 7 exercises to be performed 5 times a day at home supplemented by chewing. chewing gum 5 times a day. These last two studies nonetheless concluded the importance of carrying out other work on the subject by working on the objectives of the studies, on the tools used, and on the implementation of the exercise program.

Also, an other study cited above does not show a significant difference in mouth opening between the two rehabilitation groups, but analyzes the adhesion and shows that it is significantly higher (59 versus 41 days) in the standard rehabilitation group, less burdensome for patients. Thus, the issue of patient adherence to active rehabilitation is real and essential to take into account in studies assessing the effect of a rehabilitation program on oral opening.

The prevalence of trismus as well as its management in physiotherapy and the effectiveness of a rehabilitation program are not clearly documented in France. Our hypothesis is that currently at least 30% of patients treated by radiochemotherapy are affected by a trismus. According to national oncology nutrition guidelines, the patients most at risk for locoregional complications are those who receive oropharyngeal ≥ 54 Gray radiotherapy doses, plus concomitant chemotherapy.

It seems essential to offer these patients early and preventive management of this symptom and its consequences, throughout the duration of treatment.

This study is all the more relevant as the progress of treatment of upper aero-digestive tract cancers have allowed an improvement in survival rates, with an increase in the number of patients living with sequelae related to treatments.

The major benefit for patients will be a decrease in the loss of mouth opening during and after treatment, with the consequent improvement of the criteria of well-being and quality of life: the resumption of a normal diet, a decrease the duration of artificial nutrition, better oral hygiene, improved speech and the recovery of mimicry. All this in order to accelerate the return to the most normal social and professional life possible.

ELIGIBILITY:
Inclusion Criteria:

* Epidermoid carcinoma of the buccal cavity, oropharynx or type 1, 2 or 3 carcinoma of cavum according to the WHO classification.
* Radiotherapy (≥ 54Gy in the oropharynx) and concomitant chemotherapy (including targeted therapies) with or without surgery.
* Patients ≥ 18 years old, understanding French.
* Patients who gave their informed consent prior to the study

Exclusion Criteria:

* Disease and/or trauma with an effect on jaw mobility with permanent trismus.
* Psychiatric non-stabilized comorbidity.
* Lack of the median and lateral incisors.
* Metastatic patient.
* Legal inability or limited legal capacity.
* Medical or psychological conditions inducing incapacity of the subject to complete the study or give his/her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Trismus prevalence | 10 weeks after the end of radiochemotherapy
  The mouth opening is measured by the distance between the upper left median incisive (n°21) and the lower left median incisive (n°31) with the Therabite Range of Motion Scale. Trismus is defined as a mouth opening of less than 35mm.

CONTACTS AND LOCATIONS:
Overall Officials: kerstin faravel, Principal Investigator — Institut régional du Cancer de Montpellier
Locations (6):
- France (6):
  - ONCOGARD, Nîmes, Gard
  - CHU d'Amiens, Amiens
  - Institut Sainte catherine, Avignon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teguh DN, Levendag PC, Voet P, van der Est H, Noever I, de Kruijf W, van Rooij P, Schmitz PI, Heijmen BJ. Trismus in patients with oropharyngeal cancer: relationship with dose in structures of mastication apparatus. Head Neck. 2008 May;30(5):622-30. doi: 10.1002/hed.20760. PMID 18213726
- [Background] Rao SD, Saleh ZH, Setton J, Tam M, McBride SM, Riaz N, Deasy JO, Lee NY. Dose-volume factors correlating with trismus following chemoradiation for head and neck cancer. Acta Oncol. 2016;55(1):99-104. doi: 10.3109/0284186X.2015.1037864. Epub 2015 Apr 29. PMID 25920361
- [Background] Dijkstra PU, Huisman PM, Roodenburg JL. Criteria for trismus in head and neck oncology. Int J Oral Maxillofac Surg. 2006 Apr;35(4):337-42. doi: 10.1016/j.ijom.2005.08.001. Epub 2005 Nov 8. PMID 16280237
- [Background] Placko G, Bellot-Samson V, Brunet S, Guyot L, Richard O, Cheynet F, Chossegros C, Ouaknine M. [Normal mouth opening in the adult French population]. Rev Stomatol Chir Maxillofac. 2005 Nov;106(5):267-71. doi: 10.1016/s0035-1768(05)86038-3. French. PMID 16292219
- [Background] Cox SC, Walker DM. Establishing a normal range for mouth opening: its use in screening for oral submucous fibrosis. Br J Oral Maxillofac Surg. 1997 Feb;35(1):40-2. doi: 10.1016/s0266-4356(97)90007-3. PMID 9043002
- [Background] van der Molen L, van Rossum MA, Rasch CR, Smeele LE, Hilgers FJ. Two-year results of a prospective preventive swallowing rehabilitation trial in patients treated with chemoradiation for advanced head and neck cancer. Eur Arch Otorhinolaryngol. 2014 May;271(5):1257-70. doi: 10.1007/s00405-013-2640-8. Epub 2013 Jul 28. PMID 23892729
- [Background] van der Molen L, van Rossum MA, Burkhead LM, Smeele LE, Hilgers FJ. Functional outcomes and rehabilitation strategies in patients treated with chemoradiotherapy for advanced head and neck cancer: a systematic review. Eur Arch Otorhinolaryngol. 2009 Jun;266(6):889-900. doi: 10.1007/s00405-008-0817-3. Epub 2008 Sep 30. PMID 18825400
- [Background] Johnson J, Johansson M, Ryden A, Houltz E, Finizia C. Impact of trismus on health-related quality of life and mental health. Head Neck. 2015 Nov;37(11):1672-9. doi: 10.1002/hed.23816. Epub 2015 Jan 27. PMID 24985733
- [Background] Hogdal N, Juhl C, Aadahl M, Gluud C. Early preventive exercises versus usual care does not seem to reduce trismus in patients treated with radiotherapy for cancer in the oral cavity or oropharynx: a randomised clinical trial. Acta Oncol. 2015 Jan;54(1):80-7. doi: 10.3109/0284186X.2014.954677. Epub 2014 Sep 17. PMID 25229260
- [Background] Buchbinder D, Currivan RB, Kaplan AJ, Urken ML. Mobilization regimens for the prevention of jaw hypomobility in the radiated patient: a comparison of three techniques. J Oral Maxillofac Surg. 1993 Aug;51(8):863-7. doi: 10.1016/s0278-2391(10)80104-1. PMID 8336223
- [Background] Pauli N, Fagerberg-Mohlin B, Andrell P, Finizia C. Exercise intervention for the treatment of trismus in head and neck cancer. Acta Oncol. 2014 Apr;53(4):502-9. doi: 10.3109/0284186X.2013.837583. Epub 2013 Oct 31. PMID 24175896
- [Background] Scherpenhuizen A, van Waes AM, Janssen LM, Van Cann EM, Stegeman I. The effect of exercise therapy in head and neck cancer patients in the treatment of radiotherapy-induced trismus: A systematic review. Oral Oncol. 2015 Aug;51(8):745-50. doi: 10.1016/j.oraloncology.2015.05.001. Epub 2015 Jun 6. PMID 26058916
- [Background] French Speaking Society of Clinical Nutrition and Metabolism (SFNEP). Clinical nutrition guidelines of the French Speaking Society of Clinical Nutrition and Metabolism (SFNEP): Summary of recommendations for adults undergoing non-surgical anticancer treatment. Dig Liver Dis. 2014 Aug;46(8):667-74. doi: 10.1016/j.dld.2014.01.160. Epub 2014 May 1. PMID 24794790
- [Background] Friedman AJ, Cosby R, Boyko S, Hatton-Bauer J, Turnbull G. Effective teaching strategies and methods of delivery for patient education: a systematic review and practice guideline recommendations. J Cancer Educ. 2011 Mar;26(1):12-21. doi: 10.1007/s13187-010-0183-x. PMID 21161465
- [Derived] Faravel K, Jarlier M, Senesse P, Huteau ME, Janiszewski C, Stoebner A, Boisselier P. Response to Somay et al. Letter to the Editor Regarding "Trismus Occurrence and Link With Radiotherapy Doses in Head and Neck Cancer Patients Treated With Chemoradiotherapy". Integr Cancer Ther. 2023 Jan-Dec;22:15347354231167367. doi: 10.1177/15347354231167367. No abstract available. PMID 37038637
- [Derived] Faravel K, Jarlier M, Senesse P, Huteau ME, Janiszewski C, Stoebner A, Boisselier P. Trismus Occurrence and Link With Radiotherapy Doses in Head and Neck Cancer Patients Treated With Chemoradiotherapy. Integr Cancer Ther. 2023 Jan-Dec;22:15347354221147283. doi: 10.1177/15347354221147283. PMID 36625502